CLINICAL TRIAL: NCT03407599
Title: A Trial Comparing the Pharmacokinetic Properties of Fast-acting Insulin Aspart Between Children, Adolescents and Adults With Type 1 Diabetes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NN1218-4371; 2017-002014-31 (Registry Identifier: European Medicines Agency (EudraCT)); U1111-1197-0428 (Other: World Health Organization (WHO))
Record Dates: First submitted 2018-01-05; First posted 2018-01-23 (Actual); Last update posted 2019-06-19 (Actual); Status verified 2019-06

CONDITIONS: Diabetes; Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1 | interventions — Insulin Aspart

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Sponsor staff involved in the clinical trial is masked according to company standard procedures.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Faster aspart followed by insulin aspart (NovoRapid®) (Experimental): Participants will receive single dose of fast-acting insulin aspart followed by single dose of NovoRapid® on two separate dosing visits. The dosing visits will be separated by a wash-out period of 3-22 days.
  Interventions: Drug: Faster aspart; Drug: Insulin aspart (NovoRapid®)
- Insulin aspart (NovoRapid®) followed by faster aspart (Experimental): Participants will receive single dose of NovoRapid® followed by single dose of fast-acting insulin aspart on two separate dosing visits. The dosing visits will be separated by a wash-out period of 3-22 days.
  Interventions: Drug: Faster aspart; Drug: Insulin aspart (NovoRapid®)

INTERVENTIONS:
Drug: Faster aspart — An injection of fast-acting insulin aspart 0.2 U/kg body weight under the skin just prior to a standard meal.
Drug: Insulin aspart (NovoRapid®) — An injection of insulin aspart (NovoRapid®) 0.2 U/kg body weight under the skin just prior to a standard meal.

SUMMARY:
The study is done to compare how faster aspart is taken up, broken down and removed from the body between different age groups (children [6-11 years], adolescents [12-17 years] and adults [18-64 years]) who have diabetes. The blood sugar (glucose) lowering effect of faster aspart will also be investigated after consuming a meal replacement drink. The effects of faster aspart will be compared to the effects of NovoRapid®.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 6-64 years (both inclusive) at the time of signing informed consent
* Diagnosed with type 1 diabetes greater than or equal to 12 months prior to the day of screening
* Body mass index for children and adolescents (male and female) between the 3rd and 97th BMI percentile and for adults less than or equal to 28.0 kg/sqm

Exclusion Criteria:

* Subject who has donated any blood or plasma in the past month or more than 500 mL within 3 months prior to screening
* Smoker (defined as a subject who is smoking at least one cigarette, cigar or pipe daily)
* Not able or willing to refrain from smoking and use of nicotine substitute products during the inpatient period

Ages: 6 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 46 (Actual)
Dates: Start 2018-01-08 (Actual); Primary Completion 2018-07-05 (Actual); Study Completion 2018-07-05 (Actual)

PRIMARY OUTCOMES:
AUC(IAsp),0-12h, area under the serum insulin aspart concentration-time curve from 0 to 12 hours | 0-12 hours
  Calculated based on insulin aspart measured in blood.

SECONDARY OUTCOMES:
AUCIAsp,0-15min, area under the serum insulin aspart concentration-time curve 0 to 15 minutes | 0-15 minutes
  Calculated based on insulin aspart measured in blood.
AUCIAsp,0-30min, area under the serum insulin aspart concentration-time curve from 0 to 30 minutes | 0-30 minutes
  Calculated based on insulin aspart measured in blood.
AUCIAsp,0-1hr, area under the serum insulin aspart concentration-time curve from 0 to 1 hour | 0-1 hour
  Calculated based on insulin aspart measured in blood.
AUCIAsp,0-1½hr, area under the serum insulin aspart concentration-time curve from 0 to 1½ hour | 0-1½ hour
  Calculated based on insulin aspart measured in blood.
AUCIAsp,0-2hr, area under the serum insulin aspart concentration-time curve from 0 to 2 hours | 0-2 hours
  Calculated based on insulin aspart measured in blood.
Cmax,IAsp, maximum observed serum insulin aspart concentration | 0-12 hours
  Calculated based on insulin aspart measured in blood.
tmax,IAsp, time to maximum observed serum insulin aspart concentration | 0-12 hours
  Calculated based on insulin aspart measured in blood.
Onset of appearanceIAsp, time from trial product administration until the first time serum insulinaspart concentration greater than or equal to Lower Limit Of Quantitation (LLOQ) | 0-12 hours
  Calculated based on insulin aspart measured in blood.
Duration of exposureIAsp, time from trial product administration until the first time serum insulin aspart concentration is equal to LLOQ in the terminal part of the curve | 0-12 hours
  Calculated based on insulin aspart measured in blood.
Time to 50% Cmax, IAsp, the first time point where the insulin aspart concentration equals 50% of Cmax,IAsp | 0-12 hours
  Calculated based on insulin aspart measured in blood.
Time to late 50% Cmax,IAsp, the last time point where the insulin aspart concentration equals 50% of Cmax,IAsp | 0-12 hours
  Calculated based on insulin aspart measured in blood.
Mean change in plasma glucose concentration from 0-1 hour after administration | 0-1 hour
  Calculated based on glucose concentration measured in plasma.
Mean change in plasma glucose concentration from 0-2 hours after administration | 0-2 hours
  Calculated based on glucose concentration measured in plasma.
Mean change in plasma glucose concentration from 0-6 hours after administration | 0-6 hours
  Calculated based on glucose concentration measured in plasma.
Change from baseline in plasma glucose concentration 1 hour after administration | Pre-dose (0 hour), 1 hour
  Calculated based on glucose concentration measured in plasma.
Change from baseline in plasma glucose concentration 2 hours after administration | Pre-dose (0 hour), 2 hours
  Calculated based on glucose concentration measured in plasma.
Plasma glucose concentration 1 hour after administration | 1 hour after administration
  Calculated based on glucose concentration measured in plasma.
Plasma glucose concentration 2 hours after administration | 2 hours after administration
  Calculated based on glucose concentration measured in plasma.
Maximum plasma glucose excursion after administration | 0-6 hours
  Calculated based on glucose concentration measured in plasma.
Maximum plasma glucose concentration after administration | 0-6 hours
  Calculated based on glucose concentration measured in plasma.
Time to maximum plasma glucose concentration after administration | 0-6 hours
  Calculated based on glucose concentration measured in plasma.
Minimum plasma glucose concentration after administration | 0-6 hours
  Calculated based on glucose concentration measured in plasma.
Number of adverse events | From screening day 1 up to the study completion day 68
  Count of events
Number of hypoglycaemic episodes | From screening day 1 up to the study completion day 68
  Count of hypoglycaemic episodes

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Reporting Anchor and Disclosure (1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Hanover, Germany

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com